CLINICAL TRIAL: NCT02993029
Title: 99Tc-MDP Versus Celecoxib Treatment in Patients with Knee Osteoarthritis
Brief Title: 99Tc-MDP Treatment for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chao Ma, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: osteoarthritis
Record Dates: First submitted 2016-12-08; First posted 2016-12-14 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Treatment Outcome
Keywords: 99Tc-MDP; osteoarthritis; celecoxib
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 99Tc-MDP (Experimental): 99Tc-MDP group:15mg in 100ml normal saline intravenously dripped every twice a week for 5 weeks, every 1weeks for 10 weeks, every 2weeks for 10 weeks, every 1 month for 6 months.
  Interventions: Drug: 99Tc-MDP
- celecoxib (Active Comparator): celecoxib capsule 200mg qd by mouth.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: 99Tc-MDP — 99Tc-MDP 15mg in 100ml normal saline intravenously dripped every twice a week for 5 weeks, every 1weeks for 10 weeks, every 2weeks for 10 weeks, every 1 month for 6 months.
  Other Names: Yunke
  Arms: 99Tc-MDP
Drug: Celecoxib — Celecoxib capsule 200mg qd by mouth.
  Other Names: Xile Bao
  Arms: celecoxib

SUMMARY:
Osteoarthritis (OA) of knee is the most common form of arthritis in the world1e, and it has received growing attention in the society because of the increase of old age population, disabled people, and medical expenses from this disease. 99Tc-MDP is effective for rheumatoid arthritis. Therefore, the investigators try to investigate the effects of 99Tc-MDP treatment in patients with osteoarthritis of knee as compared with celecoxib.

DETAILED DESCRIPTION:
The prevalence of osteoarthritis of the knee (OA) is increasing worldwide and this burden will continue to increase owing to aging of the general population 99Tc-MDP is effective for rheumatoid arthritis. Consequent to an increase in incidence is the rise in the number of patients with knee OA who are prone to further deterioration of the knee. It therefore is important to better understand, control, and attempt to prevent further progression of disease in patients with knee OA. Limitations in walking, stair climbing, and squatting are common patient complaints that greatly interfere with activities of daily living and recreation. Currently there is no definite consensus on the standardized management of OA. Oral analgesic and anti-inflammatory agents are perhaps the most commonly prescribed treatments to alleviate knee OA symptoms. The failure of nonsurgical therapies to modify quality of life in knee OA patients is not surprising given their inability to alleviate physical manifestations of OA. Surgical knee OA interventions generally result in good to excellent patient outcomes. However, there are significant barriers to considering surgery, which limits clinical utility.

99Tc-MDP is actually the decay product of 99mTc-MDP (99mTc-methylene diphosphonate, a US Food and Drug Administration-approved radioactive agent widely used for bone scintigraphy). 99Tc-MDP (Chengdu Yunke Pharmaceutical, Sichuan, China) is a kind of anti-inflammatory drug patented in China (patent no. ZL94113006.1). It was approved for production by the State Food and Drug Administration of China in October 1997. 99Tc-MDP has been demonstrated to be safe and effective in the clinical treatment of immune diseases, such as rheumatoid arthritis (RA), ankylosing spondylitis (AS) and certain bone diseases, such as skeletal metastases from cancer in China. 99Tc-MDP also showed clinical effect on knee OA in our practice. Therefore, the investigators try to investigate the effects of 99Tc-MDP treatment in patients with osteoarthritis of knee as compared with celecoxib.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with painful osteoarthritis;
2. The standard uptake value (SUV) of OA related knee greater than 10 on 18F- sodium fluoride bone scan;
3. Participants voluntarily participate in the trial, and signed the informed consent.

Exclusion Criteria:

1. Knee joint replacement;
2. Inflammatory arthritis or joint infection of knee;
3. Nervous joint disease;
4. Fracture of joint;
5. Gout arthritis of the knee;
6. Traumatic arthritis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pain, stiffness and joint function of knee | baseline, and 6, 12 months after treatment.
  change of the pain, stiffness and joint function of knee (mean and standard deviation) by Western Ontario and McMaster Universities (WOMAC)Osteoarthritis Index

SECONDARY OUTCOMES:
health-related quality of life | baseline, and 6, 12 months after treatment.
  change of health-related quality of life (mean and standard deviation) by SF-36
staging of knee osteoarthritisby | baseline and 12 months after treatment.
  number of participants who have change of knee osteoarthritis staging by X-ray or CT
standard uptake value of knee | baseline and 12 months after treatment.
  change of standard uptake value (SUV,mean and standard deviation) of knee on 18F- sodium fluoride or 99Tc-MDP bone scan and change of cystic area on according CT
adverse events | 3, 6, 12 months after treatment.
  adverse events that are related to treatment

OTHER OUTCOMES:
bone mineral density | baseline and 12 months after treatment.
  The changes of bone mineral density(mean and standard deviation) in lumbar and hip by a dual energy x-ray absorotiometrv

CONTACTS AND LOCATIONS:
Overall Officials: Zhongwei Lv, MD, Principal Investigator — The 10th Hospital, Tongji University
Locations (1):
- Department of Nuclear Medicine, Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCrae F, Shouls J, Dieppe P, Watt I. Scintigraphic assessment of osteoarthritis of the knee joint. Ann Rheum Dis. 1992 Aug;51(8):938-42. doi: 10.1136/ard.51.8.938. PMID 1417117
- [Background] Lai K, Xu L, Jin C, Wu K, Tian Z, Huang C, Zhong X, Ye H. Technetium-99 conjugated with methylene diphosphonate (99Tc-MDP) inhibits experimental choroidal neovascularization in vivo and VEGF-induced cell migration and tube formation in vitro. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):5702-12. doi: 10.1167/iovs.10-6370. PMID 21666238
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Boegard T, Rudling O, Dahlstrom J, Dirksen H, Petersson IF, Jonsson K. Bone scintigraphy in chronic knee pain: comparison with magnetic resonance imaging. Ann Rheum Dis. 1999 Jan;58(1):20-6. doi: 10.1136/ard.58.1.20. PMID 10343536
- [Background] Kim HR, So Y, Moon SG, Lee IS, Lee SH. Clinical value of (99m)Tc-methylene diphosphonate (MDP) bone single photon emission computed tomography (SPECT) in patients with knee osteoarthritis. Osteoarthritis Cartilage. 2008 Feb;16(2):212-8. doi: 10.1016/j.joca.2007.05.025. Epub 2007 Jul 27. PMID 17662626
- [Background] Liu H, Guo H, Guo S, Wang J, Ye Y, Ma C. Novel treatment of 99Tc-MDP improves clinical and radiographic results for patients with osteochondral lesions of the talus. Q J Nucl Med Mol Imaging. 2019 Jun;63(2):199-206. doi: 10.23736/S1824-4785.16.02872-7. Epub 2016 Jun 21. PMID 27327630